CLINICAL TRIAL: NCT07336992
Title: Efficacy of Prophylactic Levetiracetam for Improving Functional Outcome in the Acute Phase of Intracerebral Haemorrhage: a Randomised, Double-blind, Placebo-controlled, Phase 3 Trial
Acronym: PEACH2
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 69HCL23_0934
Record Dates: First submitted 2025-09-17; First posted 2026-01-13 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2025-09

CONDITIONS: Spontaneous Intracerebral Hemorrhage
Keywords: supratentorial
MeSH Terms: interventions — Levetiracetam; Neuroimaging; Mental Status and Dementia Tests; 4-amino-4'-hydroxylaminodiphenylsulfone

STUDY DESIGN:
Intervention Model Description: This is a phase 3, national, multicentre, randomised, double-blind, 2-arm parallel-group placebo-controlled, superiority clinical trial:
  * Intervention group: Levetiracetam started within 24 hours of inclusion and continued for 1 month and 15 days.
  * Control group: Placebo started within 24 hours of inclusion and continued for 1 month and 15 days.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This is a double-blind trial. Patients and all those involved in patient management or clinical or imaging assessment of adverse events or outcomes will be masked to treatment allocation. The investigational drug will be distributed to participating centres in externally indistinguishable sealed treatment kits. Preparations of levetiracetam and placebo will be matched to ensure masking of participants and investigators, with vials, capsules, packaging, and labelling all identical in appearance.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Active Comparator): 290 patients will be recruited over 3 years in the intervention group.
  In this group, Levetiracetam should be initiated within 24 hours of randomisation. Levetiracetam (500 mg every 12 hours) will be administered intravenously for at least 48 hours and then the route of administration will be changed to oral administration at the same dosage after assessment of swallowing function. The treatment period will be 30 days at full dose, followed by a gradual tapering over 2 weeks (250 mg of levetiracetam every 12 hours for 7 days, followed by 250 mg of levetiracetam every 24 h for 7 days).
  Interventions: Drug: Treatment administration (Levetiracetam or placebo); Radiation: Neuroimaging; Diagnostic Test: National Institute of Health Stroke Scale (NIHSS); Behavioral: Modified Rankin Scale (mRS); Behavioral: Euroqol test (EQ-5D-5L); Behavioral: Montreal Cognitive Assessment (MoCA); Behavioral: Functional Assessment of Cancer Therapy - Cognitive Function (FACT-Cog); Behavioral: Hospital Anxiety and Depression Scale (HADS)
- Control Group (Placebo Comparator): 290 patients will be recruited over 3 years in the control group.
  In this group, the placebo (microcrystalline cellulose) should be initiated within 24 hours of randomisation. The placebo (500 mg every 12 hours) will be administered intravenously for at least 48 hours and then the route of administration will be changed to oral administration at the same dosage after assessment of swallowing function. The treatment period will be 30 days at full dose, followed by a gradual tapering over 2 weeks (250 mg of placebo every 12 hours for 7 days, followed by 250 mg of placebo every 24 h for 7 days).
  Interventions: Drug: Treatment administration (Levetiracetam or placebo); Radiation: Neuroimaging; Diagnostic Test: National Institute of Health Stroke Scale (NIHSS); Behavioral: Modified Rankin Scale (mRS); Behavioral: Euroqol test (EQ-5D-5L); Behavioral: Montreal Cognitive Assessment (MoCA); Behavioral: Functional Assessment of Cancer Therapy - Cognitive Function (FACT-Cog); Behavioral: Hospital Anxiety and Depression Scale (HADS)

INTERVENTIONS:
Drug: Treatment administration (Levetiracetam or placebo) — Treatment should be initiated within 24 hours of randomisation. It will be administered intravenously for at least 48 hours and then the route of administration will be changed to oral administration at the same dosage after assessment of swallowing function. The treatment period will be 30 days at full dose, followed by a gradual tapering over 2 weeks.
Radiation: Neuroimaging — Neuroimaging (brain CT or MRI) will be performed 72h post inclusion
Diagnostic Test: National Institute of Health Stroke Scale (NIHSS) — NIHSS, a clinician -reported 11-items stroke-specific severity scale, will be administered by a neurologist during all patients' study visits except at visits 1 month and 12 months.
Behavioral: Modified Rankin Scale (mRS) — This questionnaire will be administered 3 time, at inclusion, 6 months and 12 months to measure post-stroke functional status and disability
Behavioral: Euroqol test (EQ-5D-5L) — This self-reported questionnaire will be completed by patients at 6 and 12 months, to assess the multidimensional chronic consequences of stroke on their daily lives
Behavioral: Montreal Cognitive Assessment (MoCA) — This test will be administered by a neurologist at 6 months to assess patients' cognitive impairment
Behavioral: Functional Assessment of Cancer Therapy - Cognitive Function (FACT-Cog) — This self-reported questionnaire will be completed by patients at 6 months, to assess patient's cognitive function (memory, attention, concentration, language, and thinking abilities)
Behavioral: Hospital Anxiety and Depression Scale (HADS) — This questionnaire will be administered at 6 months to evaluate patients' anxiety and depression

SUMMARY:
Epileptic seizures are a common complication at the acute phase of intracerebral haemorrhage (ICH). The incidence of seizures occurring within 7 days reaches 40% when subclinical seizures are diagnosed by continuous electroencephalogram (EEG).

Some studies have suggested that early seizures are associated with haematoma expansion (Vespa., Neurology 2003), worse neurological outcomes (Gilmore., Stroke 2016) or increased mortality. By contrast, other studies have shown no association of acute seizures with long-term mortality and outcome. However, the interpretation of these works is subject to bias because almost all studies were based on clinical detection of seizures only, while it has been shown that most early seizures after ICH are clinically unrecognised and can only be diagnosed with EEG monitoring.

The PEACH trial, a double-blind, randomised, placebo-controlled, showed that clinical and/or electrographic seizures occur in more than 40% of patients with ICH and that Levetiracetam (LVT) is safe and effective in preventing these seizures. However, it remains unclear whether preventing acute seizures might lead to improved functional outcomes after ICH. An adequately powered randomised controlled trial is needed to answer whether primary seizure prophylaxis improves functional outcome in this setting. Answering this question would result in an important change in ICH acute care guidelines, which currently do not recommend primary prophylactic antiseizure treatment. As compared to research in acute ischemic stroke management, fewer clinical trials have been conducted in acute ICH and no effective medical treatments are available in this subset of patients.

The main objective of PEACH 2 is to establish if prophylactic antiseizure therapy with LVT improves functional outcome in adults with acute spontaneous ICH. Functional outcome assessed by the modified Rankin score (mRS score) six months after acute ICH will be compared between patients receiving prophylactic antiseizure therapy with levetiracetam and patients receiving placebo.

The secondary objectives are to examine the effect of prophylactic antiseizure therapy with levetiracetam versus placebo on:

* the number of early and late clinical seizures, on the short term and long term evolution of the neurologic deficit as assessed by the NIHSS, on long term functional outcome (12 months) as assessed by the mRS, on quality of life and cognitive impairment, and on haematoma expansion and mass effect on control brain imaging
* the frequency of side effects at 1 and 6 months, pneumonia at 1 month, delirium at 1 month, anxiety and depression at 1 and 6 months, and all-cause mortality at 1, 6 and 12 months.

  580 patients will be recruited over 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Spontaneous (non-traumatic) supratentorial intracerebral haemorrhage diagnosed by brain CT or MRI
* Onset of neurologic symptoms within 24 hours
* NIHSS score on admission ≤ 25
* Informed consent given by the patient or his/her legal representative
* Patients benefiting from a social insurance system or a similar system

Exclusion Criteria:

* Intracerebral haemorrhage known or suspected by study investigator to be secondary to trauma, vascular malformation, haemorrhagic transformation of ischaemic stroke, or tumour
* Current use of antiseizure drugs or history of epilepsy
* Severe renal insufficiency (creatinine clearance < 30 ml/min)
* Pregnancy or breastfeeding
* Previous history of severe depression or psychotic disorder
* Known terminal illness
* Known allergy or hypersensitivity to levetiracetam
* Known allergy or hypersensitivity to microcrystalline cellulose or lactose
* Being under legal protection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 580 (Estimated)
Dates: Start 2026-01-02 (Estimated); Primary Completion 2029-07-02 (Estimated); Study Completion 2030-01-02 (Estimated)

PRIMARY OUTCOMES:
modified Rankin Scale (mRS) score to measure the functional status (death or dependency). | 6 months after inclusion
  The mRS score will be measured by a certified neurologist, blinded to the patient study group.
  It categorises disability with reference to pre-stroke activities. mRS is a single-item scale ranging from 0 (no disability) to 5 (severe disability) and 6 (death).
  Its analysis will be performed by an ordinal logistic regression model with proportional odds and mixed effects. The treatment arm will be introduced in the model as fixed effect and the NIHSS score (≤ 15 vs >15) will be taken into account as a fixed effect. It will also take into account, as random effect, a random intercept by centre.

SECONDARY OUTCOMES:
Number of clinical seizures | within 72 hours after inclusion
Number of clinical seizures | at 1 month after inclusion
Number of clinical seizures | at 6 months after inclusion
Number of clinical seizures | at 12 months after inclusion
Change in National Institute of Health Stroke Scale (NIHSS, 11 items version) score between inclusion and 72 h, and 6 months. | At inclusion
  The NIHSS is a clinician -reported 11-items stroke-specific severity scale. This scale ranges from 0 to 42, with higher scores indicating greater severity
Change in National Institute of Health Stroke Scale (NIHSS, 11 items version) score between inclusion and 72 h, and 6 months. | At 72 hours
  The NIHSS is a clinician -reported 11-items stroke-specific severity scale. This scale ranges from 0 to 42, with higher scores indicating greater severity
Change in National Institute of Health Stroke Scale (NIHSS, 11 items version) score between inclusion and 72 h, and 6 months. | At 6 months after inclusion
  The NIHSS is a clinician -reported 11-items stroke-specific severity scale. This scale ranges from 0 to 42, with higher scores indicating greater severity
Change in modified Rankin Scale (mRS) score between inclusion and 6 months and 12 months | At inclusion
  It categorises disability with reference to pre-stroke activities. mRS is a single-item scale ranging from 0 (no disability) to 5 (severe disability) and 6 (death).
Change in modified Rankin Scale (mRS) score between inclusion and 6 months and 12 months | At 6 months after inclusion
  It categorises disability with reference to pre-stroke activities. mRS is a single-item scale ranging from 0 (no disability) to 5 (severe disability) and 6 (death).
Change in modified Rankin Scale (mRS) score between inclusion and 6 months and 12 months | At 12 months after inclusion
  It categorises disability with reference to pre-stroke activities. mRS is a single-item scale ranging from 0 (no disability) to 5 (severe disability) and 6 (death).
Score at the Euroqol (EQ-5D-5L) to assess quality of life. | At 6 months
  The EQ-5D-5L is a self-reported questionnaire composed of 5 items. The response to each item is based on a Likert scale rated from 1 (no difficulty) to 5 (inability), with a higher score reflecting worse autonomy. In addition, a question is asked about how the patients perceive their current health on a scale of 0 to 100.
  An algorithm generates scores for each domain from 0 to 100, with a score of 0 corresponding to worse health and a score of 100 corresponding to greater health.
Score at the Euroqol (EQ-5D-5L) to assess quality of life. | At 12 months after inclusion
  The EQ-5D-5L is a self-reported questionnaire composed of 5 items. The response to each item is based on a Likert scale rated from 1 (no difficulty) to 5 (inability), with a higher score reflecting worse autonomy. In addition, a question is asked about how the patients perceive their current health on a scale of 0 to 100.
  An algorithm generates scores for each domain from 0 to 100, with a score of 0 corresponding to worse health and a score of 100 corresponding to greater health.
Score at the Montreal Cognitive Assessment (MoCA) version 8.3 to assess cognitive impairment. | 6 months after inclusion
  This 30-point scale assesses visual-constructive functions, executive functions, short-term memory, attention, language, and temporo-spatial orientation. The score is pathological when it is strictly below 26/30.
Change in intracerebral haemorrhage volume (cc) | 72 hours after inclusion
  This change is defined as change in intracerebral haemorrhage volume between baseline brain imaging and control brain imaging at 72 hours
Frequency of pneumonia | 1 month after inclusion
Frequency of side effects related to treatment | 1 month after inclusion
Frequency of side effects related to treatment | 6 months after inclusion
Frequency of delirium | 1 month after inclusion
Score at the Hospital Anxiety and Depression Scale (HADS) to assess anxiety and depression | At 6 months after inclusion
  This scale has 14 items scored from 0 to 3. Seven questions relate to anxiety and seven to depression, resulting in two scores with a maximum score of 21 for each. A score of 7 or less indicates no symptomatology, 8 to 10: doubtful symptomatology, and 11 and above: definite symptomatology.
Death rate | At 1 month after inclusion
Death rate | At 6 months after inclusion
Death rate | At 12 months after inclusion
Score at the Functional Assessment of Cancer Therapy-Cognitive Function (FACT-Cog) | At 6 months after inclusion
  This scale is a self-report questionnaire composed of 37-item assesses memory, attention, concentration, language, and thinking abilities. The FACT-Cog takes into consideration the functional implications of cognitive impairment, the deficits observed by other people, the changes in cognitive function over time, and their impact on the patient's quality of life. Scoring for the FACT-Cog includes calculation of four subscales based on a 5-point Likert scale (from never/not at all (0) to several times a day/very much) : Perceived Cognitive Impairment (20 items; score range 0-80), Impact On Quality Of Life (4 items; score range 0-16), Comments From Others (4 items; score range 0-16), and Perceived Cognitive Abilities (9 items; score range 0-36). The higher the score is, the better the quality of life is.

CONTACTS AND LOCATIONS:
Overall Officials: Laurent Derex, DR, Study Director — Hospices Civils de Lyon
Locations (1):
- Hospices Civils de Lyon, Bron, France

IPD SHARING:
Plan to Share IPD: Undecided
NOT YET DECIDED